CLINICAL TRIAL: NCT01631760
Title: Identification of Plasma miRNAs as Potential Biomarkers in Asthma Exacerbation
Status: Withdrawn | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Richard Lockey, Principal Investigator, University of South Florida
Other Study IDs: Biomarkers in Asthma
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Asthma
Keywords: Asthma; Asthma Exacerbations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MicroRNA ages 5-12 yrs old: As a prospective study, we would like to look for the differential expression of microRNA in different age groups (ages 5 to 12, 13 to 55, and 56 and older) of asthma patients with exacerbation. At least 20 patients for each group is anticipated.
  Interventions: Genetic: no intervention
- MicroRNA ages 13-55 yrs old: As a prospective study, we would like to look for the differential expression of microRNA in different age groups (ages 5 to 12, 13 to 55, and 56 and older) of asthma patients with exacerbation. At least 20 patients for each group is anticipated.
  Interventions: Genetic: no intervention
- MicroRNA ages 56-85 yrs old: As a prospective study, we would like to look for the differential expression of microRNA in different age groups (ages 5 to 12, 13 to 55, and 56 and older) of asthma patients with exacerbation. At least 20 patients for each group is anticipated.
  Interventions: Genetic: no intervention

INTERVENTIONS:
Genetic: no intervention — We will be analyzing MicroRNA in subjects with Asthma Exacerbations by various age groups, Ages 5-12yrs, 13-55yrs, and 56-85yrs for genetic similarities and differences.

SUMMARY:
We hypothesize that there is a statistically significant difference in miRNA profiling and expression of subjects with asthma upon its exacerbation compared to patient's baseline level or following effective treatment of an exacerbation of asthma. Therefore, plasma miRNA profiling may provide noninvasive, highly specific and sensitive biomarkers for asthma exacerbation's detection and treatment follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Literacy: The subject must be able to read and comprehend English. Consent: The subject must have the ability to give informed consent. Type of subject: The subject must be seen in the outpatient setting at one of the clinics staffed by faculty members of the Division of Allergy and Immunology, Department of Internal Medicine, University of South Florida College of Medicine.
* Asthma: The subject must have a history of physician diagnosed asthma for at least 1 year and must have a current exacerbation of asthma requiring oral glucocorticosteroids. Asthma exacerbation is defined below.

Asthma exacerbation (relapse or de novo) is defined as either:

1. An increase of asthma symptoms (cough, wheeze, chest tightness, and /or shortness of breath) that does not resolve within 2 hours after the use of rescue albuterol or corticosteroids and requires a medical visit or
2. During a scheduled visit, the subject has acute worsening of asthma symptoms and a reduction of >20% in peak flow, which in the opinion of the investigator requires treatment with oral glucocorticosteroids.

Exclusion Criteria:

* Females who are pregnant or lactating.
* Any other coexistent lung disease (COPD, interstitial lung disease, allergic bronchopulmonary aspergillosis, TB, sarcoidosis).
* Any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the results if the condition/disease exacerbates during the study. The list of conditions/diseases that will result in exclusion if determined to be clinically significant includes, but is not limited to: uncontrolled hypertension; hematological, hepatic, neurological, thyroid, peptic ulcer, or renal disease; immunologic compromise; current malignancy.
* Past or current use of tobacco (<10 pack year smoking history and no smoking within the last 5 years).

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both genders of any racial or ethnic group, age 5-85 are eligible. The subjects should not have participated in any other experimental study in the last 30 days.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To evaluate to effect of asthma exacerbation on MiRNA profiling and expression | August 9, 2014

SECONDARY OUTCOMES:
To evaluate to effect of asthma exacerbation treatment on miRNA profiling and expression | August 2014

OTHER OUTCOMES:
To evaluate the differential expression of miRNA in different age groups ages 5 to 12, 13 to 55 and 56y and older) of asthma patients with exacerbation. | August 2014

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lockey, MD, Principal Investigator — Division of Allergy and Immunology, Department of Internal Medicine, University of South Florida College of Medicine
Locations (2):
- United States (2):
  - USF Asthma, Allergy and Immunology, Tampa, Florida
  - USF Division of Allergy and Clinical Immunology Clinical Research Unit, Tampa, Florida